CLINICAL TRIAL: NCT04388462
Title: Finite Element Analysis for Comminuted Fractures of the Midshaft of the Tibia; (Interlocking Nail +/- Blocking Screws or Locked Plating With Predicted Distribution of Locking Screws)
Brief Title: Comminuted Fractures of the Midshaft of the Tibia; (Interlocking Nail +/- Blocking Screws or Locked Plating With Predicted Distribution of Locking Screws) Choice Based on Finite Element Analysis Correlated With Clinical Outcome and Union.
Acronym: Finite Element
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sahar Ahmed Abdalbary, Associate professor, Cairo University
Other Study IDs: sahar Abdalbary; Ayman Ali Ali Saleh (Other: Cairo U)
Record Dates: First submitted 2020-05-07; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Comminuted Fracture Tibia
Keywords: Comminuted fracture, Finite element analysis, Tibia
MeSH Terms: conditions — Fractures, Comminuted | interventions — Finite Element Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- locked plating with predicted distribution of loc
  Interventions: Other: Finite element analysis
- unlocked plating with predicted distribution of loc
  Interventions: Other: Finite element analysis
- Interlocking nail +/- blocking screws
  Interventions: Other: Finite element analysis

INTERVENTIONS:
Other: Finite element analysis — Biomechanical study to describe micromotion

SUMMARY:
study is to assess the clinical and radiological results of Comminuted fractures of the midshaft of the tibia; treated with interlocking nail +/- blocking screws or locked plating with predicted distribution of locking screws, choice based on finite element analysis correlated with clinical outcome and union.

DETAILED DESCRIPTION:
FE analyses will be performed using the finite element code COSMOS/M. The three-dimensional "lower leg" FE model (LL FE model) will be used included the tibia and the fibula. The bony structures will be generated by segmentation of a data set of computed tomographies from the Visible Human Project.

Analysis of data regarding clinical outcomes and radiological assessment of healing rate and union

ELIGIBILITY:
Inclusion Criteria:

1. patients with closed comminuted fractures of the midshaft of the tibia
2. patients with age ranging from 25 to 45 years old

Exclusion Criteria:

* 1- Simple fractures of the midshaft of the tibia. 2- patients with open comminuted fractures of the midshaft of the tibia. 3- critical and ICU patients. 4- patients with ipsilateral lower limb fractures.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient with comminuted fractures of the midshaft of the tibia.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-05-02 (Actual)

PRIMARY OUTCOMES:
Healing of the fracture | 3 month
  radiographic evaluation of union rate and clinical outcomes
Tibia Pain | 3 month
  Visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Sahar, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data about the age and Phone to recall the patients. Data about Radiological investigation to be addressed by the finite element analysis